CLINICAL TRIAL: NCT00335868
Title: A Pilot Phase II Study of PHA-739358 in Patients With Chronic Myeloid Leukemia Relapsing on Gleevec or c-ABL Therapy
Brief Title: PHA-739358 in Treating Patients With Chronic Myelogenous Leukemia That Relapsed After Imatinib Mesylate or c-ABL Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald Paquette, Jonsson Comprehensive Cancer Center at UCLA
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000486219; UCLA-0601009-01; NERVIANO-AURA-6202-005
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase | interventions — danusertib

INTERVENTIONS:
Drug: danusertib
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: PHA-739358 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well PHA-739358 works in treating patients with chronic myelogenous leukemia that relapsed after imatinib mesylate or c-ABL therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Explore the clinical efficacy of PHA-739358, in terms of hematological response lasting ≥ 4 weeks, in patients with chronic myelogenous leukemia that relapsed after imatinib mesylate or c-ABL therapy.
* Explore the safety profile of this drug in these patients.
* Explore the pharmacokinetic profile of this drug and its N-oxide metabolite PHA-816359 in plasma.
* Explore the modulation of histone H3 and CRKL phosphorylation after PHA-739358 administration.
* Explore the relationship between plasma drug levels and the modulation of histone H3 and CRKL phosphorylation.
* Explore the clinical efficacy of this drug, in terms of cytogenetic response in bone marrow.
* Explore response depending on status of T315I mutation in BCR-ABL kinase.

OUTLINE: This is a pilot, open-label, multicenter study.

Patients receive PHA-739358 IV over 6 hours on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients benefitting from treatment may receive additional courses at the discretion of the investigator.

Patients undergo blood collection and bone marrow biopsies periodically for pharmacologic and biomarker correlative studies.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 16 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia confirmed by bone marrow biopsy

  * Chronic, accelerated, or blastic phase disease
* May have T315I mutation in BCR-ABL kinase
* Relapsed after prior imatinib mesylate or c-ABL therapy
* No CNS leukemia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Blood pressure ≤ 140/90 mm Hg (with or without hypertension treatment for ≥ 1 week)
* Transaminases ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No known history of HIV infection
* No active uncontrolled infection
* No grade 3 or 4 bleeding
* LVEF ≥ 45% by MUGA or ≥ 40% by transthoracic echocardiography
* No medical or psychiatric condition or laboratory abnormalities that would limit study compliance or increase risk during study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 (female) or 180 (male) days after completion of study treatment
* No significant cardiovascular disease (i.e., uncontrolled arrhythmias or unstable angina) within the past 6 months
* No major thromboembolic event within the past 6 months, including any of the following:

  * Myocardial infarction
  * Stroke
  * Transient ischemic attack
  * Pulmonary embolism
  * Noncatheter-related deep-vein thrombosis

PRIOR CONCURRENT THERAPY:

* Recovered from all acute toxic effects (excluding alopecia) of prior therapy
* More than 2 weeks since prior chemoimmunotherapy

  * Hydroxyurea must be discontinued 1 day prior to study therapy
* More than 4 weeks since prior major surgery
* No other concurrent approved or investigational anticancer treatment, including chemotherapy, biologic response modifiers, hormones, or immunotherapy
* No other concurrent investigational drugs
* No concurrent participation in another treatment clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Antileukemic response in terms of complete hematological response, no evidence of leukemia, or return to chronic phase
Overall safety profile of PHA-739358 by type, severity, timing, and relatedness of adverse events and laboratory abnormalities
Pharmacokinetics of this drug and its N-oxide metabolite PHA-816359 by measuring their plasma concentration at different times after dosing
Changes in histone H3 and CRKL phosphorylation
Correlation between changes in degree of histone H3 and CRKL phosphorylation and concurrent PHA-739358 concentrations and/or hematological response
Complete, partial, or minor cytogenetic response in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States